CLINICAL TRIAL: NCT01673659
Title: A Safety and Bioequivalence of a Mometasone Nasal Spray, 50 mcg/Actuation Compared With Nasonex® Nasal Spray 50 mcg/Actuation in the Relief of the Symptoms of Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-12-008
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test product (Experimental): Mometasone furoate 50 mcg/actuation Nasal Spray
  Interventions: Drug: Mometasone furoate
- Reference product (Active Comparator): Nasonex Nasal Spray
  Interventions: Drug: Nasonex Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): vehicle of the test product
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Mometasone furoate
  Arms: Test product
Drug: Nasonex Nasal Spray
  Arms: Reference product
Drug: Placebo nasal spray
  Arms: Placebo Nasal Spray

SUMMARY:
The objectives of this study is to demonstrate bioequivalence (comparable safety and efficacy) of the Test product to the Reference in the treatment of subjects seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Complete the informed consent/assent process.
2. Male or female between 12-65 years of age.
3. Female subjects of child-bearing potential must not be pregnant or nursing, must have a negative urine pregnancy test and abstain from sexual intercourse or use a reliable method of contraception during the study.
4. Subjects will be eligible to participate if: a) Their total rTNSS is at least 6; b) Reflective rating for "nasal congestion/stuffy nose" is a score of >2 at Visit 1; c) Reflective score of >2 for at least one (1) of the remaining three (3) allergic rhinitis symptoms.
5. A history (2 or more seasons) of seasonal allergy to at least one allergen known to be present during the study season, confirmed by a skin prick test. (A documented positive skin test within the previous 12 months is acceptable.)

Exclusion Criteria:

1. Female who is pregnant or nursing, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study.
2. Subject has a history of hypersensitivity or allergy to Mometasone, any other corticosteroids or any of the other study medication ingredients.
3. Patients who suffer from chronic signs and symptoms of Perennial Allergic Rhinitis (PAR) should be excluded from the study, unless the Investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR), rather than chronic PAR.
4. A total score of less than 6 on the rTNSS or a score less than 2 for "nasal congestion" or a score less than 2 for all of the remaining 3 symptoms.
5. Subject has any condition or abnormality of the upper airway (ex: nasal polyps, obstruction, recent nasal surgery, structural abnormality, rhinitis medicamentosa, etc.) that, in the opinion of the Investigator, could interfere with administration of the product, evaluation of the subject's condition, or other aspect of the trial.
6. Subject has experienced any upper respiratory tract infection or has experienced a sinus infection within the 30 days, or has a history of recurrent sinus infections i.e. acute or significant chronic sinusitis, preceding Visit 1.
7. Subject has a history of asthma requiring chronic treatment within two years of study start.
8. Subject lacks history of seasonal allergy to at least one allergen known to be present during the study season for at least the two preceding seasons.
9. Subject has a negative skin test for all appropriate allergens known to be present during the study season.
10. Treatment for oral Candidiasis within 30 days of starting the study, or a current oral Candidiasis infection.
11. The subject has had recent exposure (30 days) or is at risk of being exposed to chicken pox or measles.
12. Patients with any untreated fungal, bacterial, systemic viral infections within the previous 30 days.
13. Subject requires treatment with systemic corticosteroids for any condition, or has received systemic or nasal steroids within the 30 days preceding Visit 1. Hormone replacement therapy is allowed, on condition that the subject has been on a stable dosing regimen for at least 90 days and remains on the same dosing regimen during the study.
14. Subject used systemic anti-inflammatory agents* including aspirin** and non-steroidal anti-inflammatory (NSAIDs) within 3 days prior to Visit 1. (*Subjects may use Acetaminophen for pain relief, as needed, throughout the study. **Use of low-dose aspirin for cardiac prophylaxis is allowed).
15. Subject had immunotherapy (including desensitization therapy to perennial allergens or seasonal allergens not found in the current season) initiated or the subject's dosage or frequency of immunotherapy has been adjusted within the 30 days preceding Visit 1.
16. Subject had desensitization therapy to the seasonal allergen that is causing their allergic rhinitis within the previous 6 months.
17. Subject presented with conjunctivitis or any other eye signs/symptoms that are not related to the diagnosis of SAR.
18. Subject has used a topical (>1%) or ophthalmic steroid preparation within 14 days preceding Visit 1. (Topical steroid preparations used for dermatological indications are permitted in concentrations of ≤1%.)
19. Use of intranasal or systemic first generation anti-histamines, leukotriene receptor antagonists (montelukast) or other nasal decongestants within 3 days of Visit 1.
20. Use of intranasal cromolyn within 14 days of Visit 1.
21. Use of intranasal or systemic second-generation antihistamines (e.g. fexofenadine, loratadine, desloratadine, cetirizine) within 10 days of Visit 1.
22. Subject has received immune-system therapy with AIC (an investigational vaccine created using immunostimulatory sequences derived from DNA), SLIT, Oral peptide sequence at any time.
23. Subject has clinically significant acute or chronic hepatic disease.
24. Subject has a history of alcoholism, drug abuse, or problems which would likely make him/her unreliable for the study.
25. Subject has any condition or uses any medication which, in the opinion of the Investigator, might interfere with the conduct or results of the study or place the prospective subject at increased risk.
26. Subject has received tricyclic antidepressants within the 30 days preceding Visit 1.
27. Subject has been treated for attention-deficit hyperactivity disorder with an unstable dose of a methylphenidate-containing products during the 30 days preceding Visit 1, or a dose adjustment is anticipated during the study.
28. Subject or the subject's parent/legal guardian is unwilling to sign the informed consent form.
29. Subject is concurrently participating in another investigational study or using any investigational drug (or biologic) or device within the 30 days prior to Visit 1.
30. Subject plans or anticipates travel outside the allergen-rich area for more than one day during the Run-In phase (Visit 1-Visit 2), or for more than two consecutive and three total days during the Treatment Period (Visit 2-Visit 3). (Whenever possible, subjects should remain in the allergen-rich area for the 3 days preceding Visit 2 and Visit 3.)
31. Subject has a history or presence of cataracts, ocular herpes, or glaucoma.
32. Subject has a history of tuberculosis.
33. Subject has previously enrolled in this study.
34. Subject has used the Reference Product (Nasonex) within 3 months prior to Visit 1.
35. History of unresponsiveness to Mometasone Nasal Spray.
36. Members of the Investigational study staff, or family members of the Investigational study staff.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline for mean reflective Total Nasal Symptom Score (rTNSS) | 2 week treatment period

SECONDARY OUTCOMES:
Mean Change from Baseline in the mean Instantaneous Total Nasal Symptom Score (iTNSS) | 2 weeks treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States